CLINICAL TRIAL: NCT04235088
Title: Impact of Somatosensory Intensive Intervention on Motor Performance of the Upper Limb and Participation in Children With Unilateral Cerebral Palsy: a Feasibility Study
Brief Title: Impact of Somatosensory Intensive Intervention on Motor Performance in Children With Unilateral Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Jorge (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCP Somatosensory intervention
Record Dates: First submitted 2020-01-07; First posted 2020-01-21 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Unilateral Cerebral Palsy
Keywords: somatosensory intensive intervention; somatosensory processing; motor performance; participation; quality of live; occupational performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Somatosensory intensive intervention (Experimental)
  Interventions: Other: Somatosensory intensive intervention

INTERVENTIONS:
Other: Somatosensory intensive intervention — The intensive somato-sensory intervention will take place during 3 weeks, 5 days per week, for 2 hours per day (30 hours of practice). During the week-ends, some somato-sensory written activities will be explained and handed to each family (6 hours of practice) Therapy sessions will be carried out in groups and each child will have his or her own therapist in charge of his or her treatment along the whole intervention. A daily check-list, design for that purpose, will be used by the therapist in order to register the gradually increased complexity of the activities and individual progression. The principal investigator will supervise all the interventions in order to assure their uniformity, adjusting the somato-sensory training protocol to the individual needs of each subject.

SUMMARY:
This study aims to investigate the effectiveness of an intensive somatosensory intervention in the upper limb of children with hemiparesis regarding structure, function, activity and participation

Hypothesis:

Intensive somatosensory activity based intervention is effective in upper limb and hand ability in children with hemiparesis, specially regarding activity and participation

DETAILED DESCRIPTION:
Feasibility and longitudinal study with blinding of the evaluator and the person analyzing the data. The study have 4 procedures:

1. - Assessment pre-intervention
2. - Intervention: three weeks
3. - Assessment post-intervention
4. - Follow-up assessment (three months after intervention).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unilateral cerebral palsy
* Manual Ability Classification System (MACS): levels I, II y III.
* Gender: male and female
* Age: 6 to 15 years old

Exclusion Criteria:

* Existence of a moderate or severe cognitive impairment, which could interfere with the comprehension of the tester cues
* Botulinum toxic infiltration 4 months before the date of the pre-intervention assessment or during intervention or during the 3 months after the final intervention
* To have suffered any injury such as fractures and/or contusions in the upper limb in the last 12 months
* Orthopedic intervention in the 6 months preceding the study or during the study

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2020-09-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Change in Canadian Occupational Performance Measure (COPM). | baseline, immediately after intervention and follow up (3 months after intervention).
  Participation measure (family aims).
Change in Children´s hand-use Experience Questionnaire (CHEQ). | baseline, immediately after intervention and follow up (3 months after intervention).
  Activity Measure (bimanual performance).

SECONDARY OUTCOMES:
Change in Pediatric Evaluation of Disability Inventory Computer Adaptive Test (PEDI-CAT). | baseline, immediately after intervention and follow up (3 months after intervention).
  Activity measure (daily activities, mobility, social/cognitive and responsibility).
Change in Jebsen Taylor Hand Function Test. | baseline, immediately after intervention and follow up (3 months after intervention).
  Activity Measure (unimanual capacity).
Change in Box and Blocks Test. | baseline, immediately after intervention and follow up (3 months after intervention).
  Activity measure (unilateral gross manual dexterity).
Change in Sensory Profile™ 2 family Questionnaire (Winnie Dunn) | baseline, immediately after intervention and follow up (3 months after intervention).
  Evaluate a child's sensory processing patterns in the context of home, school, and community-based activities.
Change in Kidscreen Questionnaire. | baseline, immediately after intervention and follow up (3 months after intervention).
  Participation measure (Quality of live).
Change in Somatosensory Battery Assessment. | baseline, immediately after intervention and follow up (3 months after intervention).
  Body structures and functions measure. Includes: registration (Semmes Weinstein monofilaments); Two points discrimination (Aesthesiometer); Single Point Location; double simultaneous, forms stereognosis (Manual Form Perception Test_ SIPT), stereognosis of familiar objects, graphesthesia (SIPT), clinical observation of texture perception, clinical observation of proprioception, pain (algometer) and functional sensitivity (Box and Blocks without vision).
Change in Dynamometer (grip strength) | baseline, immediately after intervention and follow up (3 months after intervention).
  Body structures and functions measure (grip strength).
Change in Pinch Gauge (pinch strength). | baseline, immediately after intervention and follow up (3 months after intervention).
  Body structures and functions measure (pinch strength).

CONTACTS AND LOCATIONS:
Overall Officials: César Cuesta García, Study Director — Occupational Thinks Research Group, Autónoma University (Madrid)
Locations (1):
- Asociación para la Investigación en la Discapacidad Motriz (AIDIMO), Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No